CLINICAL TRIAL: NCT06272344
Title: Remote Programming of Cardiac Implantable Electronic Devices 2
Acronym: REACT 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2022/38
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pacemaker; Defibrillator; Telemedecine
Keywords: Implantable cardioverter defibrillator; ICD; Telemedecine; Remote monitoring; Remote programming; Cardiac implantable electronical device; Medically underserved population; Medically underserved area; Health professional shortage area
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-arm, pairwise comparison trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teleconsultation (Experimental): Teleconsultation at 6 months
  Interventions: Other: Teleconsultation

INTERVENTIONS:
Other: Teleconsultation — Teleconsultation at 6 months

SUMMARY:
Cardiac Implantable Electronic Devices (CIEDs) such as pacemakers and implantable cardioverter defibrillators need to be regularly and systematically interrogated and reprogrammed to ensure proper functioning. While remote monitoring allows for partial interrogation at a remote location, full CIED check-up and reprogramming is only possible when the patient visits a cardiologist capable of performing device programming. This can be challenging for patients and may cause unnecessary delays, particularly in settings of limited resources, enforced physical distancing, and quarantines. The aim of this study is to evaluate our previously validated remote programming solution (REACT study, NCT05366660) in outpatient device clinics which are close to the patient's home but remote from the CIED expert.

DETAILED DESCRIPTION:
Remote programming of a CIED offers multiple advantages such as shorter travel distances for the patient, reduced need for presence of specialized cardiologists and the possibility to offer expert support at remote locations or developing countries. Remote programming may be a way to mitigate disparities in health care access. The remote surveillance centre of CHU Bordeaux has previously developed and validated (REACT study, NCT05366660) a remote control system for CIED programmers that eliminates the physical presence of a cardiologist during the interrogation and programming process. The aim of this study is to evaluate this solution for the remote evaluation of CIEDs at the benefit of inhabitant of medically underserved population. Enrolled patients living >100km from the Bordeaux University Hospital will undergo there an in person evaluation of their CIED which will be compared six months later with a remote evaluation in a nurse office close to the patient's home.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both sexes over the age of 18
* Patients implanted with a cardiac pacemaker or an automatic defibrillator and an indication for device check-up (interrogation ± programming)
* Patient followed at the Bordeaux University Hospital but living more than 90km away
* Person beneficiary of social security insurance
* Informed consent confirmed in writing (at the latest on the day of inclusion and before any examination required by the research)
* Women of procreating age with effective contraception

Exclusion Criteria:

* Patients younger than 18 years old
* Patients who are incapable to understand the study design or to give informed consent.
* Pregnant or breastfeeding women
* Persons placed under legal protection
* Subject deprived of liberty on judicial or administrative decision
* Persons participating in another study who are still in their period of exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
assess the satisfaction of patients benefiting from a teleconsultation compared to a standard consultation at hospital | 6 months
  Patient satisfaction

SECONDARY OUTCOMES:
Time saving for patient | 6 months
  Time of consultation and teleconsultation
Savings on medical transport | 6 months
  Cost of medical transports for consultation and teleconsultation
Costs associated with teleconsultation | 6 months
  Global amount of costs for teleconsultation
safety of teleconsultation | 6 months
  Number of Adverse Events and technical incidents

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain MD PLOUX, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ploux S, Strik M, Varma N, Bouteiller XP, Carlier L, Lissandreau S, Ben Boujema T, Boursier D, Hugot E, Haissaguerre M, Benali K, Bordachar P. Bridging the Gap: Remote Evaluation and Programming of Cardiac Implantable Devices in Medically Underserved Areas. JACC Clin Electrophysiol. 2025 Jan;11(1):171-178. doi: 10.1016/j.jacep.2024.09.027. Epub 2024 Nov 27. PMID 39614866